CLINICAL TRIAL: NCT06038435
Title: The Effect of Cognitive Orientation Approach on Daily Occupational Performance on Executive Functions and Occupational Participation in Children With Autism Spectrum Disorder: Randomized Controlled Study With 1 Month Follow-up
Brief Title: The Effect of Cognitive Orientation Approach on Daily Occupational Performance With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Zeynep Çorakcı Yazıcıoğlu, Lecturer, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CORAKCİ-004
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Executive Function; Patient Participation
Keywords: Autism Spectrum Disorder; Cognitive Orientation; Ayres Sensory Integration
MeSH Terms: conditions — Autism Spectrum Disorder; Patient Participation; Orientation, Spatial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Orientation Approach + Ayres Sensory Integration Therapy (Experimental): Cognitive Orientation Approach on Daily Occupational Performance (CO-OP) and Ayres Sensory Integration (ASI) Therapy will be applied together
  Interventions: Behavioral: Cognitive Orientation Approach; Behavioral: Ayres Sensory Integration Therapy
- Ayres Sensory Integration Therapy Only (Active Comparator): Only Ayres Sensory Integration (ASI) Therapy will be applied
  Interventions: Behavioral: Ayres Sensory Integration Therapy

INTERVENTIONS:
Behavioral: Cognitive Orientation Approach — Cognitive training will be given for the selected occupation
  Arms: Cognitive Orientation Approach + Ayres Sensory Integration Therapy
Behavioral: Ayres Sensory Integration Therapy — Sensory integration therapy will be applied.

SUMMARY:
The goal of this clinical trial is by using the Cognitive Orientation Approach on Daily Occupational Performance, which is also supported by the literature and applied by occupational therapists, in children diagnosed with Autism Spectrum Disorder, it is aimed to determine how children's executive function scores and occupational participation change.

The main questions it aims to answer are:

* Does the Cognitive Orientation Approach on Daily Occupational Performance have an effect on executive functions?
* Does the Cognitive Orientation Approach on Daily Occupational Performance have an effect on occupational performance?

Participants will:

* Evaluations will be applied to all participants
* Divided into intervention and control groups
* The intervention group will be given "Cognitive Orientation Approach on Daily Occupational Performance" and "Ayres Sensory Integration Therapy" followed up for about 10 weeks.
* The control group will be given "Ayres Sensory Integration Therapy" followed up for about 10 weeks.
* After 10 weeks, the results between the two groups will be compared.
* After the second evaluation, both groups will be followed for 1 month and the same evaluations will be repeated.

Researchers will compare intervention and control groups to see executive functions and occupational participation.

DETAILED DESCRIPTION:
Autism spectrum disorder is a complex developmental disorder that can lead to dysfunctions in cognitive, emotion regulation, and communication skills.

At the beginning of the cognitive problems seen in children with autism, the pathophysiology in executive functions, which is affected by individual differences, comes to the fore. Difficulties related to executive functions such as cognitive flexibility and problem solving cause limitations in many basic areas, especially in daily life in autism.

The Cognitive Orientation Approach on Daily Occupational Performance, designed by Polatajko and others, is an activity-oriented problem-solving approach that uses cognitive strategies to develop motor skills in children who have difficulties during daily activities; It is a therapy method that focuses on the goal or the task itself, rather than the acquisition of functions within the activity performance. It is known that the approach is effective on social, emotional and organizational skills, especially cognitive skills in children with autism spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Autism Spectrum Disorder according to DSM-V by the Department of Child and Adolescent Mental Health
* Being between the ages of 7 years and 10 years and 11 months
* Score 30-36 points on the Childhood Autism Rating Scale
* Participation must be approved by the parent.

Exclusion Criteria:

* Having a concomitant neurological, psychiatric or orthopedic diagnosis
* Attending a program other than individual education

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
The Behavior Rating Inventory of Executive Function | 10 weeks
  It is a rating used to evaluate the behavior of children and adolescents in the home and school environment, taking into account executive functions. It is a likert scale between 1-3 points and a score between 86-258 is obtained. High score is associated with impaired executive function.
The Executive Function and Occupational Routines Scale | 10 weeks
  It evaluates children's skills such as impulsivity, verbal and non-verbal memory, self-regulation, planning and problem solving. It consists of 4 subtests including the total score. It is obtained by dividing each subtest score by the number of questions. It gives a score between 1-5 points. A high score indicates improvement.
The Short Child Occupational Profile | 10 weeks
  The profile provides a comprehensive assessment of the child's activity participation and a holistic consideration of the factors that facilitate or limit occupational participation. It consists of 7 subtests including the total score. It is a likert scale between 1-4 points. While the "environmental" subtest is between 5-20 points, the other subtests are between 4-16 points. A higher score is associated with increased occupational performance.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure | 10 weeks
  It is a person-centered approach to establishing treatment goals and assessing perceived performance and satisfaction changes over time. Performance and satisfaction subtests score between 1-5. A higher score is associated with increased occupational performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided